CLINICAL TRIAL: NCT07383662
Title: Using Students' Toolkit to Assess the Social Accountability of Dental Students at Misr International University in Egypt: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Keraa, Vice CEO Quality Assurance Unit, Misr International University
Other Study IDs: MIU-IRB-2122-157
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Social Accountability
Keywords: Social Accountability (SA); Dental school; Medical education; Dental education; Community service; Oral and Dental health equity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental students and interns

SUMMARY:
Data were collected via a paper-based questionnaire adapted from IFMSA Social Accountability Toolkit Questionnaire. The questionnaire was distributed to all students and interns during the study period, with a total of 1805 dental students and interns.

DETAILED DESCRIPTION:
A paper-based survey was conducted to assess the social accountability of the students; students from all educational years were invited to participate voluntarily. The participating students were asked to read the questions in the table (Appendix 1) carefully and rate the school's performance from 0 to 3 for each area. Then the total score was calculated by adding the scores of each question to a total and seeing where our faculty stands. Additional information on each of the questions and accompanying indicators were provided in the second column to guide students during scoring.

ELIGIBILITY:
Inclusion Criteria:

* Dental students at MIU, both males and females of different educational years and interns

Exclusion Criteria:

* Subjects who refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental students and interns at MIU
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Social accountability score | From enrollment till distribution of all questionnaires in a month
  The total score was calculated by adding the scores of each question to a total and seeing where our faculty stands. Additional information on each of the questions and accompanying indicators were provided in the second column to guide students during scoring.
  Scoring implications:
  The interpretation of the scores 0-8: Start a conversation with your classmates and school to begin to build social accountability at your school. 9-17: Your school has some social accountability strategies, look for ways to advocate to build on these existing strategies 18-26: Your school is doing well, look for areas of weakness and ways to advocate to improve social accountability. 27-36: Your school has a strong foundation in social accountability and advocates for continued growth and leadership in social accountability.

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Building Capacity in Higher Education Topic Guide 201
- [Background] Woollard B, Boelen C. Seeking impact of medical schools on health: meeting the challenges of social accountability. Med Educ. 2012 Jan;46(1):21-7. doi: 10.1111/j.1365-2923.2011.04081.x. PMID 22150193
- [Background] Alrebish SA, Taha MH, Ahmed MH, Abdalla ME. Commitment towards a better future for medical education in Saudi Arabia: the efforts of the college of medicine at Qassim University to become socially accountable. Med Educ Online. 2020 Dec;25(1):1710328. doi: 10.1080/10872981.2019.1710328. PMID 31902316
- [Background] 2. Reza Ghaffari, Ali Taghizadieh, Mozhgan Behshid , Mohammad Husein Somi, Azim Mirzazadeh, Hamid Reza Baradaran, Mark Huntington, Seyed Hasan Emami Razavi, Flora Baghban Rezvan, Fariba Salek Ranjbarzadeh. Accountability in medical education from theory to practice Tabriz 2018 statement: A step towards the implementation of this social necessity.
- [Background] 1. Boelen C., Heck J. E. (1995). Defining and measuring the social accountability of medical schools. Geneva: World Health Organization. No. WHO/HRH/95.7.